CLINICAL TRIAL: NCT04198909
Title: Optimization of a Non-invasive Electrophysiological Method for Studying the Functionality of Auditory Nerve Fibers
Acronym: ECOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratory of Neurosensory Biophysics - UMR INSERM 1107. (Unknown); Foundation of Gueules Cassées (Unknown); Region of Auvergne-Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 GIRAUDET; 2018-A02525-50 (Other: 2018-A02525-50)
Record Dates: First submitted 2019-11-28; First posted 2019-12-13 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteer; Without Hearing Disorders
Keywords: hidden hearing loss; questionnaire; hearing screening; electrocochleography
MeSH Terms: conditions — Hearing Loss, Hidden | interventions — Audiometry, Evoked Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental)
  Interventions: Diagnostic Test: Electrocochleography, electrophysiology thet for analyse the wave I generated by the auditory pathways

INTERVENTIONS:
Diagnostic Test: Electrocochleography, electrophysiology thet for analyse the wave I generated by the auditory pathways — Electrocochleography is a technique that analyses the functionality of inner ear.

SUMMARY:
Acoustic overexposure can induced temporary or hearing loss. Usually hearing loss is associated with cochlear cell damages. Recently, a new pathological entity was described and called "hidden hearing loss". In animal model, the histopathology revealed a selective reduction in the number of auditory fibers, resulting in a decrease in the amplitude of wave I of the auditory brainstem response. Electrocochleography (Ecog) is a method for recording the electrical potentials of the cochlea (e.g. wave I). In clinical routine, Ecog is performed invasively with sedation or local anesthesia. Actually, a non invasive approach could be perform but it seems necessary to optimize this method and to define reference values in healthy volunteers.

DETAILED DESCRIPTION:
The sound overexposure is a major cause of hearing disorders. The installation of hearing disorders can be temporary or permanent. Most of the time the investigators see a rise in hearing thresholds that can be accompanied by tinnitus. However, sometimes-hearing disorders aren't characterized by higher auditory threshold but by a complaint of understanding in noise. Two explanation are the either possible with a lesion at the peripheral level (sensory organ) or central lesion (auditory pathways). Peripheral damage is easily analysed by conventional tests such as the audiogram. Concerning the central lesions, through to the Electrocochleography, one sees a diminution of the wave I which corresponds to the nerve fiber injury. The wave I can more easily be analysed by the Electrocochleography method. This technique previously used an electrode deposited trans-tympanically in contact with the sensory organ. But, the evolution of a non-invasive technique is now available. However, several assemblies of the electrode are then possible without knowing the impact of these on the morphology of the wave I. Moreover, no normative values are also referenced in the literature on the population without hearing problems. It's in this context that clinical study is carried out in order to optimize the technique on the assembly of the electrode and the acoustic stimulation delivered. After this analyses and obtaining an optimal technique it's envisaged to study the morphology of the wave I in healthy volunteers aged 18-25 years. A pre-inclusion visit will verify the volunteers doesn't have a hearing disorders through a questionnaire, otoscopy, tympanometry and audiometry. Then two steps will be realized. The first is to evaluate the morphology of wave I according to assembly of electrode and acoustic stimulation delivered (machine calibration or calibration in the external auditory canal). The second step will provide normative values for people 18-25 years old who aren't hearing-impaired. Volunteers will have the choice to participate in one or both stages. The aim is to obtain wave I reference values for Electrocochleography technique. The secondary objectives are to analyse the impact of the assembly of the electrode and the adaptation of the acoustic stimulation presented.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years old
* be affiliated to a social security system
* understand (oral and written) of the French language
* be a qualified hearing with normal tympanogram and audiogram

Exclusion Criteria:

* have a complaint of hearing
* have a exposure to noise (professional and/or activities)
* refusal to participate in the study
* have ear infections and/or ENT medical history
* have cardiovascular, metabolic, neurological and psychiatric desease
* being a protected person
* healthy volunteer who has received compensation equal to or greader than 4500€ in clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 430 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Latency of wave I by electrocochleography | Day 180
  The wave I analyzed at electrocochleography will allow to obtain the latency (milliseconds) of action potential (AP)
Latency of wave I by electrocochleography | Day 360
  The wave I analyzed at electrocochleography will allow to obtain the latency (milliseconds) of action potential (AP)

SECONDARY OUTCOMES:
Hearing thresholds in decibels | Day -1 , Day 180, Day 360
  The audiometry will make it possible to obtain the hearing thresholds in decibels for all frequency of 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000, 8000, 9000, 10000, 11200, 12500 and 14000 Hz.
Acoustic reflex thresholds in decibels | Day -1 , Day 180, Day 360
  The acoustic reflex allows to evaluate the trigger threshold in decibels of the reflex for the frequencies 500, 1000, 2000, 4000Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Giraudet, Principal Investigator — Université d'Auvergne
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France